CLINICAL TRIAL: NCT01765088
Title: A Phase III Trial on Adjuvant Standard Temozolomide Chemotherapy With or Without Interferon-alpha in Newly Diagnosed High-grade Gliomas
Brief Title: A Phase III Trial on Adjuvant Temozolomide With or Without Interferon-alpha in Newly Diagnosed High-grade Gliomas
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Zhongping Chen, Professor and Chair, Department of Neurosurgery, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CSNO2012001
Record Dates: First submitted 2013-01-07; First posted 2013-01-10 (Estimated); Last update posted 2018-02-23 (Actual); Status verified 2018-02

CONDITIONS: Anaplastic Oligoastrocytoma; Anaplastic Astrocytoma; Glioblastoma
Keywords: High-grade glioma; chemotherapy; Temozolomide; Interferon-alpha
MeSH Terms: conditions — Astrocytoma; Glioblastoma; Glioma | interventions — Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- temozolomide (Active Comparator): Four weeks after radiotherapy, patients will be received 6 cycle of temozolomide (150 mg/m^2 daily on Days 1-5 of each 28 day study cycle and 200 mg/m^2 daily of subsequent cycles)
  Interventions: Drug: Temozolomide
- temozolomide +α-IFN (Experimental): Four weeks after radiotherapy, patients will be received 6 cycle of temozolomide plus α-IFN α-IFN：3mIU (3million) Day1,3,5 of each 28 day TMZ：150 mg/m^2 daily on Days 2-6 of each 28 day study cycle and 200 mg/m^2 daily of subsequent cycles
  Interventions: Drug: Temozolomide; Drug: α-IFN

INTERVENTIONS:
Drug: Temozolomide — dosed at 200 mg/m2 (150 mg/m2 for the first cycle) daily for 5 consecutive days, repeated every 28 days
  Other Names: Temodar
Drug: α-IFN — 3mIU (3million) D1，3，5
  Other Names: INTRONA
  Arms: temozolomide +α-IFN

SUMMARY:
This study is being conducted to help determine whether the addition of Interferon-alpha(α-IFN),which were determined sensitized the activity of Temozolomide(TMZ) in vivo and vitro, when given along with temozolomide during the monthly cycles that follow radiation, is able to delay tumor growth, shrink tumors, or impact how long people with newly diagnosed high-grade glioma.

DETAILED DESCRIPTION:
This study is being conducted to help determine whether the addition of Interferon-alpha(α-IFN),which were determined sensitized the activity of Temozolomide(TMZ) in vivo and vitro, when given along with temozolomide during the monthly cycles that follow radiation, is able to delay tumor growth, shrink tumors, or impact how long people with newly diagnosed high-grade glioma. Four weeks after radiotherapy, newly diagnosed WHO III-IV glioma patients will be randomised into two groups: TMZ group or TMZ+ α-IFN groups.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 years to 75 years
* newly diagnosed WHO III-IV glioma after operation and radiotherapy
* Karnofsky Performance Score ≥ 60
* Adequate bone marrow, liver and renal function
* Ability of subject to understand character and individual consequences of the clinical trial
* Written informed consent
* anticipating survival ≥2 months

Exclusion Criteria:

* Refusal to participate the study
* Known hypersensitivity or contraindication to temozolomide
* Incompletely radiation
* Pregnant or lactating females
* Malignant tumor other than brain tumor
* Contraindicated for MRI examination
* Unable to comply with the follow-up studies of this trial
* Purulent and chronic infected wounds
* Uncontrolled psychotic disorders or epilepsy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2012-09; Primary Completion 2017-12 (Actual); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Over-all survival | 5-year

SECONDARY OUTCOMES:
Quality of life | 5-year

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Guo C, Yang Q, Xu P, Deng M, Jiang T, Cai L, Li J, Sai K, Xi S, Ouyang H, Liu M, Li X, Li Z, Ni X, Cao X, Li C, Wu S, Du X, Su J, Xue X, Wang Y, Li G, Qin Z, Yang H, Zhou T, Liu J, Hu X, Wang J, Jiang X, Lin F, Zhang X, Ke C, Lv X, Lv Y, Hu W, Zeng J, Chen Z, Zhong S, Wang H, Chen Y, Zhang J, Li D, Mou Y, Chen Z. Adjuvant Temozolomide Chemotherapy With or Without Interferon Alfa Among Patients With Newly Diagnosed High-grade Gliomas: A Randomized Clinical Trial. JAMA Netw Open. 2023 Jan 3;6(1):e2253285. doi: 10.1001/jamanetworkopen.2022.53285. PMID 36705923